CLINICAL TRIAL: NCT00007904
Title: A Phase II Study Of Safety And Tolerability Of Adjuvant Chemotherapy With Continuous Infusion Paclitaxel And Dose Intense Cyclophosphamide And Hematopoietic Growth Factor Support Followed By Doxorubicin For Stage II-IIIA Breast Cancer Involving Greater Than or Equal to 10 Lymph Nodes
Brief Title: Adjuvant Stage 2-3A Breast Cancer With Positive Lymph Nodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1100; P30CA043703 (NIH); 05-00-23 (Other: University Hospitals IRB); NCI-G00-1877; CWRU1100 (Other: Case Comprehensive Cancer Center); NCI-2010-01068 (Other: NCI/CTRP)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Doxorubicin; Paclitaxel; Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A: Combination Chemotherapy (Experimental): Paclitaxel IV continuously over 72 hours on days 1-3 and cyclophosphamide IV on days 1-3. Filgrastim subcutaneously (SC) beginning on day 5 and continuing until blood counts recover or pegfilgrastim SC on day 5. Treatment repeats every 21 days for 3 courses. Then doxorubicin hydrochloride IV on day 1 and filgrastim SC beginning on day 2 and continuing until blood counts recover or pegfilgrastim SC on day 2. Treatment repeats every 21 days for 4 courses. Patients with hormone-receptor positive tumors receive oral tamoxifen citrate or oral anastrozole daily for 5 years following chemotherapy. Beginning 3-6 weeks after completion of chemotherapy, patients undergo radiation therapy 5 days a week for 6-7 weeks.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Drug: tamoxifen citrate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Neupogen (G-CSF) given at a dose of 10 ugm/kg subcutaneously starting on day 5 and continuing until ANC > 10,000/uL x1 day after the nadir cycles 1-3.
  Other Names: G-CSF, Neupogen®; recominant-methionyl human granulocyte-colony stimulating factor; granulocyte colony stimulating factor; r-methHuG-CSF
Drug: cyclophosphamide — cyclophosphamide 700 mg/m2 daily for 3 day every 3 weeks cycles 1-3
  Other Names: Cytoxan®; CTX; CPM; Neosar®
Drug: doxorubicin hydrochloride — Patients then receive doxorubicin IV on day 1.
Drug: paclitaxel — Paclitaxel 160 mg/m2 given over 72 hours by continuous infusion days 1-3
  Other Names: Taxol®
Drug: tamoxifen citrate — tamoxifen at a dose of 20 mg daily for 5 years after chemotherapy is completed
Procedure: adjuvant therapy — Patients receive paclitaxel IV continuously and cyclophosphamide IV over 2 hours on days 1-3. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until day 14 or until blood counts recover. Treatment repeats every 21 days for 3 courses. Patients then receive doxorubicin IV on day 1 and G-CSF SC on days 2-11 every 21 days for 4 courses.
Radiation: radiation therapy — Beginning 3-6 weeks after the completion of chemotherapy, patients receive radiotherapy 5 days a week for 6-7 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with filgrastim and radiation therapy works in treating patients with stage II or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of administering adjuvant paclitaxel, dose-intensive cyclophosphamide, and filgrastim (G-CSF), followed by doxorubicin and then radiotherapy in patients with stage II or IIIA breast cancer involving > 4 lymph nodes.
* Determine the incidence of febrile neutropenia in these patients during the first course of therapy.
* Compare the incidence of febrile neutropenia and duration of neutropenia in patients treated with this regimen with that seen in patients treated on protocol CWRU-4194.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Evaluate the quality of life of these patients.
* Correlate HER-2/neu overexpression with disease-free and overall survival in these patients.

OUTLINE: Patients receive paclitaxel IV continuously and cyclophosphamide IV over 2 hours on days 1-3. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until day 14 or until blood counts recover. Treatment repeats every 21 days for 3 courses. Patients then receive doxorubicin IV on day 1 and G-CSF SC on days 2-11 every 21 days for 4 courses.

Patients with hormone receptor positive disease also receive oral tamoxifen daily for 5 years beginning at the completion of chemotherapy.

Beginning 3-6 weeks after the completion of chemotherapy, patients receive radiotherapy 5 days a week for 6-7 weeks.

Quality of life is assessed days 1 and 4 of the first course of chemotherapy, day 1 of the second course, the last day of the final course, and at 6 months after the completion of treatment.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II or IIIA breast cancer

  * At least 5 axillary lymph nodes
  * No T4 or N3 disease
* No distant metastases by CT scan of the chest, abdomen, and pelvis; bone scan; and bone marrow evaluation
* No more than 8 weeks since prior lumpectomy or mastectomy with axillary node dissection

  * Negative surgical margins
* Hormone receptor status:

  * Hormone receptor status known

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No poorly controlled ischemic heart disease or congestive heart failure

Pulmonary:

* No severe chronic obstructive or restrictive pulmonary disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe diabetes mellitus
* No other severe concurrent medical or psychiatric illness that would preclude study participation
* No other malignancy within past 5 years except curatively treated ductal carcinoma in situ, lobular carcinoma in situ, or breast cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2000-07; Primary Completion 2006-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety of administering continuous infusion paclitaxel with dose intense cyclophosphamide | 9 weeks
  Paclitaxel 160 mg/m2 given over 72 hours by continuous infusion days 1-3 given concurrently with cyclophosphamide 700 mg/m2 daily for 3 day every 3 weeks cycles 1-3. Patients will be observed in the outpatient treatment area during the first 2 hours of the paclitaxel infusion for allergic reactions. Epinephrine, hydrocortisone, and IV antihistamine will be available.
To determine the incidence of febrile neutropenia with the first cycle of therapy. | 3 weeks
  A specific objective of this trial is to estimate the incidence of febrile neutropenia. The observed incidence of febrile neutropenia with the first cycle of cyclophosphamide and paclitaxel, as well as the observed number of days of grade ¾ neutropenia during the first treatment cycle, will be reported along with 95% confidence intervals.

SECONDARY OUTCOMES:
To determine days of neutrophil counts below 500/uL on this regimen during the first treatment cycle. | after 1st cycle (3 weeks)
To evaluate dose delays and dose reductions of this regimen. | at 7 cycles (21 weeks)
To determine disease-free and overall survival of this regimen. | 5 yrs after treatment
Quality of life as assessed by Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire | 6 months after treatment
  Quality of life will be assessed using the FACT-B instrument. Quality of life will be assessed at the following timepoints: Cycle 1 day 1, Cycle 1 day 4, Cycle 2 day 1, on the final day of adriamycin, and 6 months after treatment is completed.
Correlation of Her2/neu overexpression with disease-free and overall survival | 5 yrs after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brenda W. Cooper, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-LUICC, Mentor, Ohio
  - UH-Chagrin Highlands, Orange, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=cwru1100